CLINICAL TRIAL: NCT05155969
Title: Evaluating the Effect of Subanaesthetic Dose of Esketamine on Prevention of Postoperative Depression in Patients Undergoing Cardiac Surgery：a Randomized, Double-blind, Placebo-controlled Pilot and Feasibility Trial
Brief Title: Intravenous Esketamine on Prevention of Postoperative Depression in Patients Undergoing Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anshi Wu (Other)
Responsible Party: Sponsor-Investigator, Anshi Wu, Head of Anesthesiology, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10110815
Record Dates: First submitted 2021-12-08; First posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Postoperative Depression
Keywords: esketamine; postoperative depression; cardic surgey
MeSH Terms: interventions — Esketamine; Ketamine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eskatamine group (Experimental): Low-dose esketamine (0.3 mg/kg in 100 ml normal saline) is intravenously infused in 40 minutes before anesthesia induction
  Interventions: Drug: Esketamine
- Placebo group (Placebo Comparator): Placebo (40 ml normal saline) is intravenously infused in 40 minutes before anesthesia induction.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Esketamine — esketamine (0.3 mg/kg in 100 ml normal saline) is intravenously infused 40 minutes before anesthesia induction
  Other Names: Ketamine hydrochloride
  Arms: Eskatamine group
Drug: Normal saline — Normal saline will be administrated intravenously at the dural opening, with a total dose of 0.5 ml/kg and continual infusion for 40 minutes.
  Other Names: saline
  Arms: Placebo group

SUMMARY:
Esketamine is a general anesthetic with anti-depressant effects at subanaesthetic doses. This study hypothesized that intraoperative administration of ketamine would prevent or mitigate postoperative depressive symptoms in surgical patients.

DETAILED DESCRIPTION:
Single subanaesthetic doses of i.v. esketamine may significantly improve symptoms in psychiatric patients with major depression.

In patients undergoing cardiac surgery, postoperative depressive symptoms are common.

This study hypothesizes that low-dose esketamine has a preventive effect on postoperative depression. However, evidence in this aspect is insufficient. The purpose of this study is to investigate the effect of a subanaesthetic dose of ketamine on POD for patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1:Patients scheduled for heart surgery
* 2:Moderate to severe depressive symptom measured by the qualified psychiatric doctors
* 3:Over 18 years of age
* 4:American Society of Anesthesiologists physical status I-III

Exclusion Criteria:

* 1:History of epilepsy
* 2:Major depression disorder patients undergoing antidepressive therapy within 2 weeks
* 3: Psychiatric illness
* 4: Drug abuse
* 5:History of allergy to esketamine
* 6:Hyperthyroidism
* 7:Patients can not cooperate with investigators on psychiatric assessments
* 8:Pregnant or breastfeeding woman
* 9:refuse to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Response rate | Postoperative 5 Days
  ≥50% reduction in MADRS scores from the baseline value. The MADRS is a 10-item tool, with scores ranging from 0 to 60, and determining the severity of depression

SECONDARY OUTCOMES:
Anxiety symptom | Postoperative 5 days
  The anxious symptom is defined as a GAD-7 score no less than 10. The GAD-7 is a 7-item tool, with scores ranging from 0 to 21, The higher the score, the worse the anxiety.
Postoperative delirium | 1-7days after surgery, on the 30th day after surgery
  Postoperative delirium will be assessed by the Confusion Assessment Method for the Intensive Care Unit Scale (CAM-ICU)
Postoperative insomnia | Postoperative 5 days
  Postoperative insomnia is defined as an ISI score of no less than 15. ISI is a 7-item tool, with scores ranging from 0 to 28, The higher the score, the worse insomnia.
Severe pain | Postoperative 3 days.
  The incidence of severe pain within first postoperative three days, which is defined as mean and peak numerical rating scale (NRS) are higher than 5.
Postoperative 30-day quality of life reported by SF-36 | postoperative 30 days
  The quality of life will be evaluated by the 36-Item Short-Form Health Survey, SF-36 at postoperative 30 days SF-36 is a 36-item tool, with scores ranging from 1 to 100, The higher the score, the better the quality of life.
Postoperative complications include psychiatric symptoms evaluated by Brief Psychiatric Rating Scale (BPRS) | Postoperative 5 days
  Postoperative complications
Psychiatric manic symptoms assessed through the 11-item Young Mania Rating Scale (YMRS) | Postoperative 5 days
Psychiatric dissociative symptoms measured by the Clinician-Administered Dissociative States Scale (CADSS). | Postoperative 5 days
Postoperative pain | Postoperative 2 days
  The postoperative pain will be evaluated by Numerical pain scale（NRS） NRS is a tool with scores ranging from 1 to 10, the higher the score, the more intense the pain

CONTACTS AND LOCATIONS:
Overall Officials: Anshi Wu Wu, Ph.D, Study Chair — Beijing Chao-Yang Hospital, Capital Medical Unive
Locations (2):
- China (2):
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Beijing, Beijing Municipality